CLINICAL TRIAL: NCT06454084
Title: Investigation of Endothelium-dependent Vasodilation in Human Gingiva Depending on Serum Estrogen Level
Brief Title: Investigation of Endothelium-dependent Vasodilation in Human Gingiva
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Semmelweis University (Other)
Responsible Party: Principal Investigator, Dr. Vag Janos, professor, Semmelweis University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2023/2025
Record Dates: First submitted 2024-06-06; First posted 2024-06-12 (Actual); Last update posted 2024-06-12 (Actual); Status verified 2024-06

CONDITIONS: Vasodilation; Oral Soft Tissue Conditions
Keywords: spreading vasodilation; gingival microcirculation; LSCI
MeSH Terms: conditions — Aneurysm | interventions — Acetylcholine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Acetylcholine 0,1 mg/mL and 1 mg/mL and 10 mg/mL (Experimental): Vasodilator solution is dropped on the labial surface of the lateral incisor, which penetrates into the gingival sulcus.
  In the dose-response study, 0,1 mg/mL, 1 mg/mL, and 10 mg/mL acetylcholine solution is dropped into the gingival sulcus, and every solution remains there for 2:30 minutes between them is always a 30-second long pause.
  In the second phase of the study, where the sex differences are monitored, 10 mg/mL acetylcholine solution is dropped into the gingival sulcus for 15 minutes
  Interventions: Drug: Acetylcholine Chloride

INTERVENTIONS:
Drug: Acetylcholine Chloride — Vasodilator solution

SUMMARY:
The first aim of this study is to create a cumulative dose-response curve for acetylcholine in men (low serum estrogen levels) to determine the lowest concentration with which we can induce a maximal vasodilation effect on the human gingiva. Furthermore, the second aim of this study is the characterization of the age-dependent effect of sex hormones on gingival blood flow, as well as of the gender differences by applying this concentration to premenopausal men and women with low and high estrogen levels, as well as to postmenopausal subjects.

DETAILED DESCRIPTION:
Gender differences were observed in studies according to gingival microcirculation between physiological circumstances and during wound healing as well.

For blood flow measurement, Laser Speckle Contrast Imaging is a reliable tool. It has good reproducibility, does not touch the measured surface, is easy to use, and can simultaneously measure on a bigger surface.

Two wells are fabricated on the surface of the right lateral incisor (test site) and the labial surface of the left central incisor (control site). These wells are opened towards the high-permeability gingival sulcus, so the dropped solutions acetylcholine vs. physiological saline can easily penetrate the gingival tissues. After applying the solutions, the blood flow is monitored for 19 minutes.

In the study's second phase, blood sampling is taken before the gingival blood flow measurement.

ELIGIBILITY:
Inclusion Criteria:

* healthy systemic and periodontal conditions

Exclusion Criteria:

* systemic disease and medication
* periodontal disease
* smoking

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — women and men
Enrollment: 80 (Estimated)
Dates: Start 2023-09-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
1. Blood flow change after applying the test solution | 19 minutes
  The change in blood flow will be measured after applying the test solution

CONTACTS AND LOCATIONS:
Locations (1):
- Department for Restorative Dentistry and Endodontics, Semmelweis University, Budapest, Hungary